# INFORMED CONSENT FORM FOR PARTICIPATION IN A CLINICAL TRIAL AND CONSENT DECLARATION

# for an adult patient capable of giving consent personally

version 1.0, 06/03/2024

TITLE: One Step Nucleic Acid Amplification (OSNA) versus ultrastaging to detect sentinel lymph node metastasis in endometrial cancer: a randomized, multicenter, controlled trial (SENT-OSNA study).

U.O.C. Gynecologic Oncology

Principal Investigator: Prof. Francesco Fanfani

Phone: 06 3015 3421

# Dear Sir/Madam,

The information contained in the following information sheet is very detailed. We ask you to agree to participate in the trial ONLY after carefully reading this sheet and having an IN-DEPTH DISCUSSION with a member of the research team who will dedicate the NECESSARY TIME to ensure that you fully understand what is being proposed.

It is your right to be informed about the purpose and characteristics of the trial so that you can make an informed and free decision about whether to participate.

This document aims to inform you about the nature of the trial, its purpose, what participation will entail for you, including your rights and responsibilities.

We encourage you to carefully read the following information. The researchers involved in this project, listed at the beginning of this document, are available to answer any questions you may have. No question that comes to mind is trivial: do not hesitate to ask it!

In addition to discussing with us, you may also talk about the proposal in this document with your family doctor, your relatives, and other people you trust. Take all the time you need to decide. You can take an unsigned copy of this document home to reflect on it or discuss it with others before making a decision. If you choose not to participate in the trial, you will still receive the best possible care for your condition/disease.

Your refusal will not be interpreted as a lack of trust in any way.

# **The Principal Investigator**

#### INFORMED CONSENT FORM

Dear Madam/Sir,

At the A. Gemelli University Hospital Foundation-IRCCS, a study titled "Single-phase amplification of nucleic acids (OSNA) versus ultrastaging for identifying metastases in sentinel lymph nodes in patients with endometrial cancer: a randomized, multicenter, controlled study (SENT-OSNA study)" is being conducted. This research is international and multicenter, meaning it involves several hospitals and care centers in Italy and other European countries.

To carry out this research, we would like to collaborate with and seek the participation of individuals who, like you, meet the scientific criteria for the evaluation that will be conducted. Whether you decide to participate in this study or not will have no impact on the care you receive, and the doctors will continue to follow you with the utmost attention.

Before deciding whether to accept or refuse participation, we kindly ask you to read these pages carefully, taking all the time you need, and to ask for clarification if anything is unclear or if you require further details. Additionally, if you wish, you may seek advice from your family members or trusted doctor before making a decision.

#### WHAT THE STUDY AIMS TO DO

The general objective of the study is to compare the effectiveness of two different methods: the OSNA (One Step Nucleic Acid Amplification) method versus ultrastaging, in identifying metastases in sentinel lymph nodes of patients with endometrial carcinoma.

Sentinel lymph node mapping (SLN) is widely used in the staging process of endometrial carcinoma. The status of the sentinel lymph nodes is an important prognostic factor and provides critical information for the proper treatment of this condition.

#### WHAT THE STUDY INVOLVES

As per clinical practice, all patients must undergo pre-operative evaluation, which includes hysteroscopic biopsy, transvaginal ultrasound, abdominal magnetic resonance imaging, and/or computed tomography (to be performed within 60 days of the surgical procedure).

The investigator's design includes a pre-operative randomization of patients enrolled in this study to determine whether sentinel lymph node analysis should be performed using the OSNA method or the ultrastaging method. The term "randomized" means that the assignment to one of the above-mentioned treatment groups will be random, and will not be influenced by the physician or the subject's condition.

# WHAT YOUR PARTICIPATION IN THE STUDY INVOLVES

Your participation in the study requires that you undergo the standard surgical treatment currently recommended in the most recent national and international guidelines: total hysterectomy, bilateral salpingo-ophorectomy, sentinel lymph node mapping, or alternatively pelvic lymphadenectomy.

The sentinel lymph nodes used in this study will be dissected following the routine surgical procedure and will be analyzed via ultrastaging or OSNA.

The surgical approach may be laparoscopic or robot-assisted depending on your body mass index, determined by your weight and height.

The study involves a 4-year patient recruitment period and 3 years of follow-up, for a total of 7 years. A total of 1,922 patients with the same disease as yours will participate in this research.

Participation in the study will not incur any additional costs for you, nor will any compensation be provided.

#### WHAT ARE THE RISKS OF PARTICIPATING IN THE STUDY

This study aims to explore the sensitivity and specificity of OSNA in identifying lymph node metastases, comparing it to the existing standard (lymph node ultrastaging).

The OSNA device is CE-marked and has been demonstrated to be intrinsically safe and reliable in various types of cancers, including endometrial cancer.

#### WHAT BENEFITS WILL YOU RECEIVE BY PARTICIPATING IN THE STUDY

No direct benefits are expected for you from participating in this study, but your participation will allow us to gather additional information about the disease you are affected by.

#### STUDY RESULTS AND CONFIDENTIALITY OF COLLECTED INFORMATION

All of your data will be pseudo-anonymized, meaning that a code will be assigned to you that is not directly traceable to your identity, and the data will be recorded electronically. This code will not allow your identification outside the medical treatment center.

Regarding the processing of personal data, you will refer to the specific information provided for consent to the processing of personal data, which will be handed to you separately on another sheet.

# WHAT HAPPENS IF YOU DECIDE NOT TO PARTICIPATE IN THE STUDY – POSSIBLE ALTERNATIVE TREAT-MENTS

You are free to choose not to participate in the study. In this case, you will still receive all the standard therapies and treatments available for your condition, without any penalties, and the doctors will continue to provide the necessary care and attention.

#### WHAT HAPPENS IN CASE OF DAMAGE

An institutional insurance policy covers this study.

# **DISCONTINUATION OF THE STUDY**

Your participation in this research program is entirely voluntary, and you may withdraw from the study at any time by informing the Principal Investigator. In this case, the data collected up to the time of withdrawal will be considered in aggregate and anonymous form for the final analysis.

Likewise, the study may be discontinued if:

- 1. The physician does not observe any benefit or if unwanted effects or other issues arise.
- 2. New information becomes available and continuing the study is no longer in your best interest.
- 3. You do not follow the agreed-upon rules for participating in the study.
- 4. You become pregnant during the study.
- 5. The study is terminated by the involved authorities or the sponsor.

In these cases, you will be promptly informed about further treatments available for your disease, and you can discuss this with your doctor. The center will continue to provide the necessary care and attention.

If new data become available that may influence your decision to continue in the study, you will be promptly informed. If you decide to continue in the study, you may be asked to sign a new informed consent form highlighting the update.

#### INFORMATION ABOUT THE STUDY RESULTS

If you request it, at the end of the study, the overall results of the study, and particularly those related to your participation, will be communicated to you.

#### ADDITIONAL INFORMATION

For further information and communications during the study, you can contact the following staff:

- Prof. Francesco Fanfani (06 3015 3452) francesco.fanfani@policlinicogemelli.it
- Prof. Giovanni Scambia
- Dr. Nicolò Bizzarri
- Dr. Maria Consiglia Giuliano
- Dr. Giuseppe Parisi

The research protocol that has been proposed to you has been reviewed and approved by the CET Lazio Area 3. The CET has, among other things, verified the compliance of the study with Good Clinical Practice Guidelines and the ethical principles expressed in the Declaration of Helsinki, ensuring that your safety, rights, and well-being are protected.

If you consider it appropriate to report any events or issues related to the study you have participated in to individuals not directly involved in the study, you can contact the CET that approved the study (Ethical Committee Lazio Area 3).

# WHO ORGANIZES AND SPONSORS THIS STUDY?

The study is promoted and funded by the A. Gemelli University Hospital Foundation under the leadership of Prof. Francesco Fanfani.

We thank you for the attention and time you have dedicated to reading and discussing this document.

If you decide to participate in the study, you will be provided with a copy of this Information Sheet and a Consent Form to sign and keep.

# **INFORMED CONSENT FORM**

(This declaration must be signed and dated by both the patient and the physician who conducted the informed consent discussion.)

| I DECLARE |
|---|
| ☐ I have received thorough explanations from Dr regard- |
| ing the request to participate in the research study, as outlined in the information section, and I was pro- |
| vided with a copy of this document, which is part of this consent, on |
| ☐ I have been clearly informed and I understand the nature, objectives, procedures, expected benefits, po- |
| tential risks, and inconveniences, as well as alternative treatment options to the proposed clinical trial. |
| ☐ I have had the opportunity to ask any questions to the study investigator, and I have received satisfac- |
| tory answers. |
| ☐ I have had sufficient time to reflect on the information provided. |
| a thave had sufficient time to reflect on the information provided. |
| ☐ I have had enough time to discuss the information with others. |
| ☐ I have been informed that the study protocol and all related documents have been approved by the rele- |
| vant Ethical Committee. |
| ☐ I am aware that the research may be stopped at any time. |
| ☐ I have been informed that I will be updated on any new information that could affect the safety of the |
| research, and that for any issues or additional questions, I can contact the principal investigator or their col- |
| laborators. |
| ☐ For the best protection of my health, I understand the importance of informing my general practitioner |
| about my participation in this study. |
| , production of the second of |
| ☐ I am aware of the importance of providing all relevant information (medications, side effects, etc.) to the |
| study investigator. |
| ☐ I have been informed that the results of the study will be shared with the scientific community, protect- |
| ing my identity in accordance with privacy laws. |
| ☐ I am aware that any decision expressed in this consent form can be revoked at any time and without jus- |
| tification. |
| tineation. |
| ☐ I have received a copy of this consent form. |
| Location and Date: |
| Dationtle Name (Drinted). |
| Patient's Name (Printed): |
| Patient's Signature: |

| (If the patient is unable to read or sign, an independent witness must be present during the entire informed consent discussion. The witness must personally sign and date the informed consent form after the form and any other written information have been read and explained to the subject, and the subject has given verbal consent to participate in the study.) |
|---|
| In this case: |
| I, the undersigned, |
| ject, having had the opportunity to ask any questions they deemed necessary, freely agreed to participate in the study. |
| Date Independent Witness Signature |
| Date Signature of the Physician Providing the Information |

# **DOCTOR'S DECLARATION OF CONSENT COLLECTION**

| Location and Date: Name and Surname (printed) of the doctor who provided the information and collected the consent: Signature (and stamp) |
|---|
| ☐ I have provided the patient with information on how the results of the study will be communicated to them. |
| ☐ I have not exerted any coercion or undue influence in requesting this consent; |
| $\Box$ I have clearly explained the possibility of withdrawing from the study at any time or modifying any decisions made; |
| ☐ I have given the Patient sufficient time and the opportunity to ask questions regarding the study; |
| ☐ I have verified that the Patient has sufficiently understood the information provided to them; |
| I also declare that: I have provided the Patient with thorough explanations regarding the aims of the study, the procedures the potential risks and benefits, and possible alternatives; |
| that the Patient has voluntarily consented to participate in the study. |
| DECLARE |
| in my capacity as: □ Principal Investigator □ Delegated Investigator |
| I, the undersigned (FIRST NAME - LAST NAME), |

This form is an integral part of the informed consent process and must be kept together with the informed consent information sheet.



(Art. 13 e 14 del GDPR EU 2016/679)

Study Promoter: The Agostino Gemelli University Hospital Foundation IRCCS

(hereinafter referred to as "Foundation")

Largo Francesco Vito, n. 1 - 00168 - Roma

Name of the study:

One Step Nucleic Acid Amplification (OSNA) versus ultrastaging to

detect sentinel lymph node metastasis in endometrial cancer: a randomized, multicenter, controlled trial (SENT-OSNA study).

**Principal Investigator** Prof. Francesco Fanfani

UOC Ginecologia Oncologica Policlinico Agostino Gemelli IRCCS

Rome ITALY

Version 1.0, 06/03/2024

The Agostino Gemelli University Hospital Foundation IRCCS (hereinafter referred to as "Foundation") as the Data Controller:

- In accordance with the responsibilities outlined in the Good Clinical Practice regulations (D.L. 211/2003);
- In compliance with the provisions:
  - ✓ Of EU Regulation 2016/679 of the European Parliament and Council regarding the protection of natural persons with regard to the processing of personal data, and the free movement of such data (hereinafter GDPR EU 2016/679);
  - ✓ Of Legislative Decree no. 196 of June 30, 2003, as amended by Legislative Decree no. 101 of August 10, 2018;
  - ✓ Of the Authority's provision concerning the processing of special categories of data, pursuant to Article 21, paragraph 1, of Legislative Decree no. 101 of August 10, 2018;
  - ✓ Of the Garante's resolution on the "Guidelines for the processing of personal data in the context of clinical trials of medicinal products" of July 24, 2008, and subsequent amendments,

will process personal data to achieve the objective of the study.

REV.: 03/04/2023 Pag. 1 di 6



(Art. 13 e 14 del GDPR EU 2016/679)

DATA CONTROLLER (Article 13, paragraph 1, letter a of the GDPR) The Promoter's contact details are as follows:

- Largo Francesco Vito, no. 1 00168 Rome
- Tel. +39 06 30151
- PEC: protocollo.generale.gemelli@pec.it

# DATA PROTECTION OFFICER (DPO) (Article 13, paragraph 1, letter b of the GDPR)

The Data Protection Officer (DPO), designated by the Data Controller pursuant to Article 37 of the GDPR, can be contacted by addressing correspondence to the Data Controller's office or by emailing: dpo@policlinicogemelli.it and at the PEC address: dpo.gemelli@pec.it. However, it should be noted that the Promoter will process only pseudonymized data of the enrolled subjects.

# LEGAL BASIS AND PURPOSE OF THE PROCESSING (Article 13, paragraph 1, letter c of the GDPR)

Personal data (any information related to an identified or identifiable natural person), including data concerning special categories (Article 9 of the GDPR) related to health status, will be processed upon obtaining consent, as the legal basis for processing according to Articles 6, paragraph 1, letter a) and Article 9, paragraph 2, letter a) of the GDPR. Specifically, the aforementioned data will be processed for the following purposes:

| Medical research, including clinical trials of medicinal products, conducted based on a project that has received a reasoned favorable opinion from the competent Ethics Committee (prospective/interventional study); |
|---|
| Conducting a study using data previously collected for healthcare purposes or for the execution of prior research projects, or projects derived from biological samples previously collected for health protection purposes, subject to a reasoned favorable opinion from the competent Ethics Committee (retrospective/observational study); |
| Scientific and statistical research aimed at safeguarding public health in the medical, biomedical, and epidemiological fields, survey (prospective observational); |
| The establishment, integration, and/or maintenance of a Registry, as per the title of the study indicated on page 1. |

DATA PROVISION (Article 13, paragraph 1, letter e of the GDPR)

REV.: 03/04/2023 Pag. 2 di 6



(Art. 13 e 14 del GDPR EU 2016/679)

Participation in the Study is voluntary and requires the provision of consent. Therefore, failure to consent to the processing of data for the purpose of participating in the project will prevent enrollment.

The data may be communicated between entities acting as independent Data Controllers within the Study for the purposes stated above, to the extent that they play the role of participating center and the communication of data is essential for conducting the Study itself. Personal data will not be disclosed, except in anonymous and/or aggregated form, in such a way that it cannot be traced back to any individual subject.

As required by the clinical trial regulations, your data may also be transmitted to the Ethics Committee and the competent authorities, in a manner that ensures confidentiality.

In accordance with Article 3 of the Ministry of Health Decree of November 30, 2021, and Law No. 3/2018 (Lorenzin Law), the data related to the Study and its results may be transferred for registration purposes, with or without profit, to another Promoter who will fully take over the ownership of personal data processing related to the trial, following the procedures set forth by the referenced ministerial decree and after the transmission of the relevant documentation to AIFA (Italian Medicines Agency) and the competent Ethics Committee.

If necessary for the purposes of the study, data may be transferred to third countries outside the European Union. In such cases, the transfer will occur in compliance with the rules of Chapter V of the GDPR (Articles 44 and following), ensuring an adequate level of protection of personal data, established contractually, including through specific clauses.

# **FUTURE RESEARCH (Article 5, paragraph 1, letter b) of the GDPR)**

In accordance with Article 5, paragraph 1, letter b) and Recital 33 of the GDPR, data subjects can provide specific consent for further use of their personal data for future research activities concerning the same condition addressed in the study, as long as these activities are compatible with the purposes for which the data were originally collected.

Consent for future research is voluntary and therefore, refusal to consent will not affect participation in the current study or the care provided.

# DATA PROCESSING METHODS (Article 13, paragraph 1, letter f of the GDPR)

Data processing will involve a series of operations (collection, recording, storage, consultation, and modification of personal data, etc.) using manual and computer-based tools, strictly related to the purposes for which the data were collected, ensuring that security, confidentiality, integrity, and availability of the data are maintained at every stage of processing.

REV.: 03/04/2023 Pag. 3 di 6



(Art. 13 e 14 del GDPR EU 2016/679)

While ensuring the adoption of technical and organizational measures to guarantee an adequate level of security, specific technical measures and precautions will be implemented to increase the security of the data processed for the execution of the study. Data access will be controlled through appropriate authentication and authorization systems, based on the roles and access needs of the personnel involved in the processing. Additionally, pseudonymization techniques and other solutions will be used to ensure the data cannot be directly attributed to any specific individual.

Data collected by the Clinical Trial Center will be identified by an alphanumeric code, which will replace the participant's name, so that only the physician and authorized personnel can associate this code with the participant's name (pseudonymization).

The data will be processed exclusively by authorized personnel who are subject to professional secrecy and the legal obligation of confidentiality, respecting the protection of the rights and dignity of the data subject.

Within the Study, your data may be processed with the cooperation of entities appointed as "Data Processors" (external entities processing data on behalf of the Data Controller), in compliance with the provisions of Article 28 of the GDPR.

# STORAGE (Article 13, paragraph 2, letter a of the GDPR)

The data provided will be stored for a period no longer than necessary to achieve the purposes for which they were processed, and in any case, for 25 years in accordance with Article 58 of EU Regulation No. 536/2014 from the completion of the study. At the end of this period, the data will be deleted.

# **EXERCISE OF RIGHTS (Article 13, paragraph 2, letter b of the GDPR)**

Pursuant to Articles 15, 16, 17, 18, and 21 of GDPR EU 2016/679, the data subject:

- a) has the right to request from the Data Controller access to personal data, rectification, supplementation, deletion, restriction of processing of data concerning them, or to object to the processing of such data where the conditions set forth in the GDPR apply;
- b) has the right to file a complaint with the Data Protection Authority, following the procedures and guidelines published on the official website of the Authority: <a href="https://www.garanteprivacy.it">www.garanteprivacy.it</a>.

The data subject may exercise the above rights at any time by contacting the Data Controller and their Data Protection Officer at the contact details provided in this notice.

The Data Controller undertakes to communicate to the data subject any necessary changes in the processing of personal data carried out for the purposes described above. The data subject may, at any time and without providing any justification, withdraw their consent and discontinue their participation in the study. In this case, no further data will be collected concerning them, with the

REV.: 03/04/2023 Pag. 4 di 6



(Art. 13 e 14 del GDPR EU 2016/679)

exception of the use of any data already collected to determine, without altering it, the results of the research. The withdrawal of consent does not affect the lawfulness of the processing based on consent before its withdrawal.

# RIGHT TO FILE A COMPLAINT WITH THE SUPERVISORY AUTHORITY (Article 13, paragraph 2, letter d of the GDPR)

Pursuant to Article 77 of the GDPR and without prejudice to any other administrative or judicial remedy, if the data subject believes that the processing concerning them violates the Regulation, they have the right to file a complaint with the competent supervisory authority, which is the Data Protection Authority, as per Article 153 of Legislative Decree 196/03 as amended by Legislative Decree 101/18, following the procedures described on the institutional website <a href="https://www.gpdp.it">www.gpdp.it</a>.

# Consent to the Processing of Data for Scientific Research Purposes for Adults Pursuant to Article 7 of the GDPR

Having acknowledged the information provided pursuant to Article 13 of the GDPR, of which this form is an integral part:

| The undersigned |
|---|
| First Name: Last Name: |
| Tax Code: Tel: |
| As the Data Subject: |
| □ gives consent □ denies consent |
| to the processing of data for research purposes, as outlined in the information notice. |
| □ gives consent □ denies consent |
| to the processing of data for the establishment, integration, and/or maintenance of the Registry. |
| □ gives consent □ denies consent |
| to the processing of data for future research purposes within the limits specified in the information notice. |
| notice. |
| □ gives consent □ denies consent |
| for the results of analyses and any unexpected findings emerging during the experimental activities to be communicated to: |
| □ Myself |

REV.: 03/04/2023 Pag. 5 di 6



(Art. 13 e 14 del GDPR EU 2016/679)

| □ Family member (Last Name and First Name | ) Contact: |
|-----------------------------------------------|------------|
| <del></del> | |
| ☐ Cohabitant/spouse (Last Name and First Name | ) Contact: |
| <del></del> | |
| □ Family doctor (Last Name and First Name | ) Contact: |
| Signature of the Data Subject | |

REV.: 03/04/2023 Pag. 6 di 6